CLINICAL TRIAL: NCT01499381
Title: Evaluation of a Novel Circulating Microvesicle-Based Multi-analyte Assay for the Detection of Prostate Cancer in Men With Elevated Risk for Prostate Cancer; the EMBRACE1 Study
Brief Title: EMBRACE1: Prostate Biorepository
Status: Completed | Type: Observational
Sponsor: Caris Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRMDA-0001-1011
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine prostate biopsy patients

SUMMARY:
The objective of this multi-center prospective observational clinical study is to evaluate the clinical performance of the Carisome Prostate assay as an aid in the diagnosis of prostate cancer in men that have been scheduled for a prostate biopsy. Primarily, results of the Carisome Prostate assay will be compared with pathology results of prostate biopsy procedures. Secondarily, the performance of the Carisome Prostate test will be compared to the current standard of care for the detection of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men scheduled for a routine prostate biopsy expected to produce a pathology evaluation and report
* Blood draw within 7 days prior to scheduled prostate biopsy procedure
* Blood draw on the day of but prior to biopsy

Exclusion Criteria:

* Any previous diagnosis of cancer with the exception of non-melanoma skin cancer
* Any prior or ongoing treatment for prostate cancer including prostatectomy or hormone therapy
* Prostate biopsy within one month of blood draw
* Previous enrollment in the Caris Life Sciences Biorepository

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men scheduled for routine prostate biopsy
Sampling Method: Probability Sample
Enrollment: 1290 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Carisome Prostate Assay with prostate biopsy outcome | up to 6 months
  Association of Carisome Prostate Assay result with prostate biopsy outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Caris Science, Inc., Phoenix, Arizona, United States